CLINICAL TRIAL: NCT03601962
Title: Evaluate the Effects of Aqualief® Mucoadhesive Tablets (a Food Supplement Based on Carnosine and Hibiscus) in Patients Who Developed Oral Xerostomia as Consequence of Radiotherapy for Head and Neck Cancer
Brief Title: Effects of Aqualief® in Patients With Xerostomia as Consequence of Radiotherapy for Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrolment rate
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Latis S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HF07-16-31
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Xerostomia; Asialia; Hyposalivation; Mouth Dryness
Keywords: Xerostomia; pH; Saliva; Aqualief; Carnosine; hibiscus; oral health
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo controlled, cross over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aqualief® tablets (Experimental): oral mucoadesive tablets
  Interventions: Dietary Supplement: Aqualief
- Placebo tablets (Placebo Comparator): oral mucoadesive tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Aqualief — 400mg oral mucoadesive tablets
  Arms: Aqualief® tablets
Other: Placebo — 400mg Placebo oral mucoadesive tablets
  Arms: Placebo tablets

SUMMARY:
The treatment of xerostomia is aimed to increase existing saliva flow or replace lost secretions, the control of the state of oral health, the control of dental caries, and the treatment of possible infections.

Therapy options in xerostomia depend on the presence of residual secretion or the absence of it. When residual secretory capacity is present, it is advisable to regularly stimulate the salivary glands by mechanical or gustatory stimuli as supportive oral care.

Aqualief® is a food supplement based on carnosine and hibiscus. These two ingredients are mixed in specific proportions to form a pH buffering system which maintains the pH of the oral cavity at the proper value which is required for the regular secretion of saliva.

DETAILED DESCRIPTION:
Xerostomia is the biggest and chronic side effect of the RT for head and neck cancer. To treat xerostomia different approach should be followed at the same time: to increase existing saliva flow or replace lost secretions, to control the state of oral health, to control dental caries and to treat possible infections18.

When residual secretory capacity is present, it is advisable to regularly stimulate the salivary glands by mechanical or gustatory stimuli as supportive oral care.

The salivary flow can be stimulated by the use of sugarless chewing gum or xylitol/sorbitol candy or through parasympathomimetic drug such as pilocarpine. Pilocarpine is a natural alkaloid that activates cholinergic receptors, authorized to treat xerostomia. Due to its main mechanism of action, pilocarpine has some muscarinic side effects19, especially vomiting, sweating, headache, increased urinary frequency, wheezing, watery eyes, nausea and gastrointestinal intolerance, hypotension, rhinitis, diarrhea, and visual disturbances. Pilocarpine has also some use restrictions that make it not prescribable to certain patients (patients with asthma, high blood pressure, heart diseases and in therapy with β-blockers cannot use pilocarpine because this drug is a nonselective antagonist of muscarinic receptors and, therefore, it can interfere with the cardiac and respiratory functions).

Acupuncture seems to alleviate radio-induced xerostomia but it mechanism of action is not totally clear and systematic reviews indicate its efficacy as doubtful20,21.

Other products are under investigation and their efficacy in xerostomia due to RT is still unclear.

Aqualief® is a food supplement based on carnosine and hibiscus. These two ingredients are mixed in specific proportions to form a pH buffering system which maintains the pH of the oral cavity at the proper value which is required for the regular secretion of saliva.

Aqualief® is designed as a mucoadesive tablet that will adhere to the cheek internal side, to have a prolonged action. It is expected to gradually release the ingredients over a period of at least two hours.

Aqualief® is being tested in a clinical study on 70 subjects with grade 1-2 xerostomy enrolled at the Dental Clinic of the University of Insubria. The study is currently ongoing therefore results are not yet available.

The aim of this clinical study is to evaluate if Aqualief® can be efficacious in the increasing of the saliva production in patients suffering for xerostomia as consequence of previous RT for head and neck cancer.

To this purpose, this double blind cross over study has been designed: 100 patients will be treated for 8 days with Aqualief®/placebo and then, following a 10 days wash-out period, for further 8 days with placebo /Aqualief®.

ELIGIBILITY:
Inclusion Criteria:

* Male and female which are 18 years of age or older
* Patients willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures
* Subjects presenting:hyposalivation of grade 2 or greater (according to CTCAE scale vers. 4) and an objective, unstimulated salivary flow between 0.1 and 0.25 ml/min following radiation or radiation + systemic therapies with curative intent (definitive or postoperative), for tumors located in the head / neck region, completed from at least 6 months and free from cancer disease
* Absence of infections in the oral cavity
* Absence of antibiotics and antifungal treatments or any odontoiatric procedure in the 10 days before each treatment phase of the study.

Exclusion Criteria:

* Contraindications in administration of carnosine and hibiscus
* Known hypersensitivity to the components present in the product.
* Subjects taking products or medications to reduce symptoms of salivary gland hypofunction (Pilocarpine etc.)
* Patients with other underlying conditions that can cause xerostomia.
* Use of experimental drugs within 30 days prior to enrollment or during the study.
* Presence of clinical conditions that may interfere with the study evaluations.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Saliva Production | Change from baseline to 8 days of treatment
  Change of saliva production, without mechanical stimulation.

SECONDARY OUTCOMES:
pH of the mouth cavity evaluation | Change from baseline to 8 days of treatment
  Change of oral pH
Xerostomia Evaluation (XQ-I questionnaire) | Change from baseline to 8 days of treatment
  Change of xerostomia following treatment
MD Anderson Dysphagia Inventory (MDADI) questionnaire | Change from baseline to 8 days of treatment
  Change of Dysphagia following treatment
Adherence to the treatment by accountability | Total tablets used from baseline to 8 days of treatment
  Accountability of used/unused tablets
Patient's global satisfaction | from baseline to 8 days of treatment
  Report from patients the facility to use and palatability of the product

CONTACTS AND LOCATIONS:
Overall Officials: Ester Orlandi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy